CLINICAL TRIAL: NCT01452204
Title: Pulsed Electromagnetic Field in Patients With Impingement Shoulder: A Randomized, Placebo-Controlled Clinical Trial
Brief Title: Pulsed Electromagnetic Field (PEMF) in Impingement Shoulder
Acronym: PEMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Diego Galace de Freitas, MSc Student Diego Freitas, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEMF01
Record Dates: First submitted 2011-09-19; First posted 2011-10-14 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2011-10

CONDITIONS: Impingement Shoulder
Keywords: PEMF; magneto; shoulder; impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed Electromagnetical Field (Experimental)
  Interventions: Other: Pulsed Electromagnetical Field and Exercise
- Placebo (Placebo Comparator)
  Interventions: Other: Pulsed Electromagnetical Field and Exercise

INTERVENTIONS:
Other: Pulsed Electromagnetical Field and Exercise — G1: MT, three times per week lasting 30' each session. G2: placebo MT, 3 X week lasting 30'each session. After 3 weeks of application of MT, will begin a program of exercises.
  Other Names: PEMF; Pulsed Electromagnetical Field; Exercise

SUMMARY:
In the past many authors have reported the abnormal contact between the rotator cuff and coracoacromial arch, but the exact etiology was not clearly understood. Thus, the objectives of this study relate specifically to improve the symptoms and rehabilitation of shoulder function of the patient:

1. Assess the effectiveness of magnet therapy in the treatment of impingement of the rotator cuff;
2. Assess whether the application of magnetic therapy 3 times a week for three weeks, may be effective as a single treatment of impingement of the rotator cuff;
3. Assess whether the combination of magnetic therapy with therapeutic exercises is more effective than magnetic therapy only;
4. Evaluate the benefits of magnetic therapy associated with therapeutic exercise in the short and long term.
5. Assess the effectiveness of the modulation of pulsed electromagnetic field at 25 Hz and 20 mT in patients with shoulder impingement syndrome.

DETAILED DESCRIPTION:
1. Randomization of the patients 1.1) Duration of wash-out Having made the proper screening of patients undergoing the study, all pre-selected patients should discontinue any medications that might influence the symptoms of impingement syndrome (such as analgesics, antiinflammatory, chondroprotective, etc.) for a period of 7 days.

   1.2) Randomization

   The investigators have chosen a total sample of 30 patients undergoing the study. Only one will be treated the shoulders of patients, if there are cases of bilateral impingement syndrome (IS). Patients will be equally distributed in two groups, receiving first place:

   Group 1: treatment with magnetic therapy, three times per week lasting 30 minutes each session.

   Group 2: placebo of magnet therapy (MT), three times per week lasting 30 minutes each session.

   Randomization will be done as follows: initially 10 patients will be selected to be evaluated by a blinded evaluator and by the end of the evaluation, the patient will randomly choose a paper folded into 2 parts, which will be inside a plastic bag. Inside this bag there will be 10 paper folded in the same way and with the same color and size, where in three of them will say "A", two of them written in "B", three of them written in "C" and two of them "D" . Patients were drawn papers written "A" and "D" will be selected for group 1 and patients to raffle papers written "B" and "C" will be selected for group 2. After the drawing paper, the same can not be placed back in the bag. Randomization will be done this way so that all patients can also be divided into two groups and for the blind assessor does not know which group the patient was allocated.
2. PLAN OF STUDY 2.1) Assessment 1: Patients selected for study are those referred to our outpatient musculoskeletal physiotherapy with a diagnosis of impingement syndrome grade II and grade III. All will be evaluated by a blinded investigator, who uses the Visual Analogue Scale (VAS), the rating scale of Constant and University of California, Los Angeles (UCLA) shoulder rating scale, and measurement of rotator cuff muscle force (external and internal rotation) and shoulder elevation.

2.2) Assessment 2: After 3 weeks of treatment only with the applications of magneto therapy, a new assessment will be equal to an evaluation made by an assessor blinded, who do not know which patients are exposed to placebo or not. After the third evaluation, all patients will continue with the sessions of magnetic therapy (placebo or not), but now associated with specific therapeutic exercises for the treatment of impingement syndrome of the shoulder. The assessment consists of two re-evaluation of all parameters previously in an evaluation.

2.3) Evaluation 3: The third evaluation will happen after three weeks of treatment with magnetic therapy and exercises over again a blind assessor will evaluate patients in the same manner as in evaluation 1 and 2. After this evaluation, patients receive high treatment and receive a booklet of exercises to help them to practice proper exercises for the shoulder at home.

2.4) Evaluation 4: The fourth review will occur six months after the third evaluation, where the main objective is to evaluate the efficacy of treatment without the guidance of a physiotherapist and without weekly applications of magnetic therapy.

* Application of methods: The investigators have chosen a total sample of 30 patients undergoing the study. Only one will be treated the shoulders of patients, if there are cases of bilateral impingement syndrome. Patients will be equally distributed in two groups, receiving first place: Group 1: treatment with magnetic therapy, three times per week lasting 30 minutes each session. Group 2: placebo of magnet therapy, three times per week lasting 30 minutes each session.After the first 3 weeks of application of magnetic therapy, will begin a program of therapeutic exercises (kinesiotherapy) equally to all patients in both groups. These exercises will be conducted after each application of magnetic therapy and all patients will receive a brochure guiding them to perform exercises at home. The applications of magnetic therapy will continue to be 3 times per week with 30 minutes duration each application, but this time associated with exercise, treatment will be done for another 4 weeks. After these four weeks, patients will be reassessed by the scale of Constant and UCLA to evaluate the overall function of the shoulders that received placebo treatment and the magneto.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have a diagnosis of impingement of the rotator cuff grade II or grade III. For patients with grade III, they must present at least 90 ° of active elevation of the affected shoulder-free. Patients with extensive lesions of the rotator cuff will be deleted.
2. The patient must be aged between 30 and 50 years, of both sexes.
3. Patients should not use any anti-inflammatory, analgesic and / or chondroprotective by at least one week before the start of treatment.
4. The patient must not have been subjected to intra-articular injection of corticosteroids for at least 30 days before the start of treatment.
5. The patient can not be being subjected to physical therapy for at least 30 days before the start of treatment.
6. Patient must have at least 3 months of discomfort and / or symptoms of impingement syndrome.

Exclusion Criteria:

1. Make use of systemic anti-inflammatory medications and / or topics during the study.
2. Patient presenting during pregnancy or postpartum.
3. A patient with cancer, even if you are treated.
4. Having been subjected to surgery on the shoulder to receive the study treatment
5. submit inflammatory joint diseases (such as rheumatoid arthritis, lupus, gout, etc.) except for the impingement of the rotator cuff.
6. Patients who do not submit high active-free up to 90 degrees (minimum) of the affected shoulder will be deleted. These cases are specific to patients with extensive lesions of the rotator cuff and have no function of this muscle group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rotator cuff muscle force | 3 weeks after exercise
  Patients selected are those referred with a diagnosis of impingement syndrome grade II and III. All will be evaluated by a blinded investigator, who uses measurement of rotator cuff muscle force after 3 weeks of exercise treatment.

SECONDARY OUTCOMES:
Rotator cuff muscle force | 3 months post-exercise follow up
  Patients selected are those referred with a diagnosis of impingement syndrome grade II and III. All will be evaluated by a blinded investigator, who uses the measurement of rotator cuff muscle force

CONTACTS AND LOCATIONS:
Overall Officials: Diego DG Galace, Study Chair, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Galace de Freitas D, Marcondes FB, Monteiro RL, Rosa SG, Maria de Moraes Barros Fucs P, Fukuda TY. Pulsed electromagnetic field and exercises in patients with shoulder impingement syndrome: a randomized, double-blind, placebo-controlled clinical trial. Arch Phys Med Rehabil. 2014 Feb;95(2):345-52. doi: 10.1016/j.apmr.2013.09.022. Epub 2013 Oct 15. PMID 24139986